

#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Multiparametric MRI and MRE Assessment of Liver Fibrosis in patients treated for HCC 2016-1113

| Subtitle: Patient Consent | integrande (and the contraction of the contraction |
|---|---|
| Study Chair: Priya Bhosale | |
| Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB - a committee that reviews research studies).

#### STUDY SUMMARY

The goal of this clinical research study is to collect additional imaging information in patients with liver cancer who will receive treatment outside of the study. This study is for patients who are already receiving standard-of-care MRIs to have another similar type of imaging called MRE (Magnetic resonance elastography) for research purposes. Researchers want to learn if MRE scanning can make it easier to see if the treatment is working, and some newer types of MR imaging such as T1W Dixon and other advanced techniques may be included to also help with seeing if the treatment is working.

This is an investigational study. MRE is FDA approved and commercially available methods to check the status of liver scarring. Using MRI with MRE scanning techniques in patients with liver cancer is investigational.

The doctor can explain how MRE is designed to work, as well as T1W Dixon and other advanced techniques if applicable.

Future patients may benefit from what is learned in the study. There are no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment. If you take part in this study, you may experience side effects.

You can read a list of potential side effects below in the Possible Risks section of this consent.

Your active participation in this study will be over after the last MRE scan is complete.

You and/or your insurance provider will be responsible for the costs of the standard-of-care MRI and CT scan. The MREs and CT images of the thighs that are done for this study will be performed at no cost to you.

You may choose not to take part in this study. You may still have your routine MRIs without taking part in this study.

#### 1. STUDY DETAILS

If you agree to take part in this study, you will have a standard-of-care MRI followed by an MRE scan for research purposes before you start your planned treatment and after 12 weeks (+/- 2 weeks) of treatment. Having an MRE performed may add up to 30 minutes to your normal scan time, for a total time of 30-90 minutes on the MRI table each time. Mayo Clinic will receive images from your MRE scan for processing. AMRA Medical Inc. will receive images and will use their software to measure fat in the soft tissue and muscle. If your doctor orders a CT scan before or after your MRI scan, the CT images may be sent to AMRA for comparison with the MRI images. The images sent to Mayo Clinic and AMRA will not have identifying information that could link to your personal information.

For 5 patients, CT scans of the thighs will be added to your normal CT scan if not already scheduled at baseline, at 3-6 months after your planned treatment, and then if at any time the disease gets worse. The study staff will let you know if this applies to you.

Information will also be collected from your medical record, such as your age, height, weight, ethnicity, and type of treatment, and the results of blood tests and liver biopsies you have had.

Information from your medical records will be continued to be reviewed for up to 5 more years.

Up to 50 participants will be enrolled in this study (up to 45 patients with cancer and up to 5 healthy volunteers who will also have an MRI for research purposes). All will take part at MD Anderson.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The known side effects are listed in this form, but they will vary from person to person.

During the **MRI/MRE**, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some people, especially those who tend to feel uncomfortable in small or closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI/MRE staff and the scanning will be stopped if you wish. The MRI/MRE will require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent. This may cause skin irritation, bleeding, and/or infection. You may have an allergic reaction to the contrast agent.

The magnetic field used in MRI/MRE scanning may harm you if you have certain types of metal in your body (as might be found in pacemakers, neurostimulators, or certain clips). It may cause problems with devices, such as pacemakers. If you have metal in your body or devices such as a pacemaker, you should discuss this with the study doctor.

Taking part in this study can result in risks to an unborn baby, so you should not have an MRE scan while pregnant. If you are pregnant, your doctor may recommend that you have another exam, or postpone the MRE scan.

CT scans send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. When a CT scan of the abdominal area is taken, material may be inserted into the rectum to better define the bowel. You will usually drink liquid to help define various abdominal organs. This may cause nausea and/or vomiting. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study.

This study may involve unpredictable risks to the participants.

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson or Diagnostic Imaging Clinical Research Committee for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

### **Additional Information**

- 4. You may ask the study chair (Dr. Priya Bhosale, at 713-792-0221) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. If you withdraw from this study, you can still

choose to be treated at MD Anderson. If you withdraw from the study, the study staff may ask if they can continue collecting the results of routine care from your medical record.

- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, Diagnostic Imaging Clinical Research Committee, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- This study is sponsored and/or supported by: Diagnostic Imaging Clinical Research Committee.

#### **Future Research**

Your personal information is being collected as part of this study. This information, or data, may be used by researchers at MD Anderson or shared with other researchers and/or institutions for use in future research.

Before being shared for future research, every effort will be made to remove your identifying information from any data. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data are used for future research. If this research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data.

Your personal information is being collected as part of this study. This data may be used by researchers at MD Anderson or shared with other researchers and/or institutions for use in future research.

If you do not want your data to be used for future research, tell the study doctor. You may withdraw your participation at any time by telling your study team. If you decide to withdraw, the data and test results already collected from your scheduled procedures from routine medical care will be kept and may be used.

## <u>Authorization for Use and Disclosure of Protected Health Information (PHI):</u>

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Diagnostic Imaging Clinical Research Committee, who is a sponsor or supporter of this study, and/or any future sponsors/supporters of the study
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

Mayo clinic will receive 3D Magnetic Resonance Elastography (MRE) images for post-processing analysis. AMRA Medical Inc. will receive images and will use their software to measure fat in the soft tissue and muscle. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study; only the study investigators will have access to this data.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.

Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.

- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the

| consent form for this study, or have had it read to me. I have about it, ask questions, and talk about it with others as nee permission to enroll me on this study. By signing this cons any of my legal rights. I will be given a signed copy of this | ded. I give the study chair ent form, I am not giving up |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| PRINTED NAME OF PARTICIPANT | |
| WITNESS TO CONSENT I was present during the explanation of the research to be part 2016-1113. | performed under Protocol |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY A witness signature is only required for vulnerable adult participants. | DATE CHAIR) |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSE | NT |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant ar representative, using language that is understandable and have fully informed this participant of the nature of this student and risks and that the participant understood this explanation | appropriate. I believe that I ly and its possible benefits |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |

| <u>IRANSLATUR</u> | | |
|---|---|---|
| subtractions) into | | it additions or<br>isted the people |
| • | ne of Language)<br>t by translating all questions and<br>pant. | I responses during the |
| NAME OF TRANSLATOR | SIGNATURE OF TRANSLATOR | DATE |
| ☐ Please check here if the translator was a member of the research team. (If checked, a witness, other than the translator, must sign the witness line below.) | | |
| SIGNATURE OF WITNESS TO<br>(OTHER THAN TRANSLATOR<br>OR STUDY CHAIR) | THE VERBAL TRANSLATION<br>, PARENT/GUARDIAN, | DATE |
| PRINTED NAME OF WITNESS | TO THE VERBAL TRANSLATI | ON |